CLINICAL TRIAL: NCT07266012
Title: Incorporating the Venous Excess Ultrasound Score (VExUS Score) Into Contemporary Haemodynamic Risk Assessment in Pulmonary Arterial Hypertension: The INVEXUS-PAH Study
Acronym: INVEXUS-PAH
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sahra Asena Balcioglu, Resident Physician, Cardiology Department, Istanbul University - Cerrahpasa
Other Study IDs: 2025/618IUCIC
Record Dates: First submitted 2025-11-23; First posted 2025-12-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Arterial Hypertension (PAH); Pulmonary Arterial Hypertension (PAH) (WHO Group 1 PH)
Keywords: VExUS; Pulmonary Arterial Hypertension; Risk Stratification; Venous Congestion; Right Ventricular Function; doppler ultrasound
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PAH Cohort: Adults with World Health Organization (WHO) Group 1 pulmonary arterial hypertension undergoing non-invasive assessment with the Venous Excess Ultrasound Score (VEXUS) and the ESC/ERS 2022 simplified four-strata risk model during routine clinical follow-up. No intervention is administered; this is an observational cohort with a single study visit in which VEXUS, 6MWT, BNP, WHO-FC and recent haemodynamic parameters are collected.

SUMMARY:
This prospective observational study aims to evaluate the relationship between the Venous Excess Ultrasound Score (VEXUS) and the ESC/ERS 2022 simplified four-strata risk assessment model in adult patients with World Health Organization (WHO) Group 1 pulmonary arterial hypertension (PAH). The study investigates whether VEXUS can enhance risk stratification and predict haemodynamic congestion by correlating VEXUS with functional, biochemical, and invasive haemodynamic parameters.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a progressive disorder characterised by increased pulmonary vascular resistance, right ventricular overload, systemic venous congestion, and high mortality. The ESC/ERS 2022 simplified four-strata model (low, intermediate-low, intermediate-high, high risk) guides treatment decisions using WHO functional class, 6-minute walk distance, and BNP/NT-proBNP levels.

However, biochemical markers may be costly or insufficiently sensitive to early haemodynamic deterioration.

VEXUS (Venous Excess Ultrasound Score), a point-of-care ultrasonographic method assessing hepatic, portal, and renal venous Doppler patterns, has shown promise in representing venous congestion.

This study evaluates whether VEXUS correlates with ESC/ERS risk categories and invasive haemodynamic parameters including right atrial pressure, mean pulmonary arterial pressure, pulmonary vascular resistance, cardiac output, and pulmonary output. The study further aims to explore whether integrating VEXUS into PAH follow-up may strengthen risk assessment.

ELIGIBILITY:
Inclusion Criteria

* Adults aged ≥18 years
* Established diagnosis of WHO Group 1 pulmonary arterial hypertension (PAH)
* Stable outpatient clinical status at the time of VExUS ultrasonography
* Venous Excess Ultrasound Score (VExUS) evaluation performed with adequate ultrasonographic acoustic windows
* Clinically indicated right heart catheterisation (RHC) performed within ±60 days of VExUS assessment
* Availability of ESC/ERS 2022 simplified risk assessment variables (WHO functional class, BNP/NT-proBNP, and 6-minute walk distance)
* Ability to provide written informed consent

Exclusion Criteria

* Pulmonary hypertension other than WHO Group 1, including:

  * PH due to left heart disease (WHO Group 2)
  * PH due to chronic lung disease or hypoxaemia (WHO Group 3)
  * Chronic thromboembolic pulmonary hypertension (CTEPH; WHO Group 4)
  * Multifactorial PH (WHO Group 5)
  * Eisenmenger syndrome
  * Complex or unrepaired congenital heart disease
* Suspected pulmonary veno-occlusive disease (PVOD)
* Pulmonary capillary haemangiomatosis (PCH)
* Acute decompensated right heart failure
* Severe renal dysfunction (eGFR <30 mL/min/1.73 m²)
* Severe hepatic impairment (Child-Pugh Class C)
* Congestive hepatopathy
* Active infection
* Pregnancy
* Inability or unwillingness to provide informed consent
* Poor ultrasonographic acoustic window preventing adequate VExUS scoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with World Health Organization (WHO) Group 1 pulmonary arterial hypertension (PAH) who are being followed at a tertiary pulmonary hypertension centre. Participants represent a real-world cohort of clinically stable PAH patients attending routine outpatient follow-up visits. All participants undergo non-invasive assessment including VEXUS ultrasonography, 6-minute walk test (6MWT), WHO functional class evaluation, and BNP measurement at the study visit. Recent right and/or left heart catheterisation data (performed within ±2 months for standard clinical indications) are collected from medical records. Patients with other forms of pulmonary hypertension, Eisenmenger syndrome, pulmonary veno-occlusive disease, or pulmonary capillary haemangiomatosis are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Correlation Between the VExUS Score and Invasive Haemodynamic Parameters | At the single study visit (Day 0)
  Correlation between the VExUS Score (0-3 Doppler-based venous congestion score) and invasive haemodynamic measurements obtained by right heart catheterisation, including pulmonary vascular resistance (PVR; Wood units), right atrial pressure (RAP; mmHg), Fick-derived cardiac output (L/min) and pulmonary blood flow (PBF; L/min).

SECONDARY OUTCOMES:
Correlation Between the VExUS Score and Non-Invasive Clinical Markers | Day 0
  Correlation between the VExUS Score and serum B-type natriuretic peptide (BNP; pg/mL), WHO functional class (4-level ordinal scale) and six-minute walk distance (metres), which form key components of current ESC/ERS risk stratification models.
Correlation Between the VExUS Score and Echocardiographic RV-PA Coupling Indices | Day 0
  Correlation between the VExUS Score and tricuspid annular plane systolic excursion (TAPSE; mm) and the TAPSE/systolic pulmonary artery pressure ratio (unitless).
Predictive Value of the VExUS Score for Elevated Pulmonary Vascular Resistance (≥ 6 Wood Units) | Day 0
  Evaluation of the predictive performance of the VExUS Score for identifying patients with elevated pulmonary vascular resistance (≥ 6 Wood units). Predictive metrics (including odds ratios) will be reported.
Incremental Contribution of the VExUS Score to ESC/ERS Four-Strata Risk Classification | Day 0
  Change in ESC/ERS simplified four-strata risk category after incorporation of the VExUS Score, including net reclassification and risk-category shifts.

CONTACTS AND LOCATIONS:
Overall Officials: SAHRA ASENA BALCIOGLU, MD, Principal Investigator — ISTANBUL UNIVERSITY-CERRAHPASA INSTITUTE OF CARDIOLOGY
Locations (1):
- Istanbul University-Cerrahpasa Institute of Cardiology, Istanbul, FATIH, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified individual participant data (IPD) related to primary and secondary outcome measures may be shared with qualified researchers upon reasonable request. No direct identifiers or protected health information will be released.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 12 months after publication of the primary manuscript and for up to 3 years thereafter.
Access Criteria: Requests must be submitted in writing to the principal investigator. Data will be provided only for methodologically sound proposals and after review by the institutional data governance committee. A data use agreement (DUA) will be required.

REFERENCES:
- [Result] Beaubien-Souligny W, Rola P, Haycock K, Bouchard J, Lamarche Y, Spiegel R, Denault AY. Quantifying systemic congestion with Point-Of-Care ultrasound: development of the venous excess ultrasound grading system. Ultrasound J. 2020 Apr 9;12(1):16. doi: 10.1186/s13089-020-00163-w. PMID 32270297
- [Result] Boucly A, Weatherald J, Savale L, Jais X, Cottin V, Prevot G, Picard F, de Groote P, Jevnikar M, Bergot E, Chaouat A, Chabanne C, Bourdin A, Parent F, Montani D, Simonneau G, Humbert M, Sitbon O. Risk assessment, prognosis and guideline implementation in pulmonary arterial hypertension. Eur Respir J. 2017 Aug 3;50(2):1700889. doi: 10.1183/13993003.00889-2017. Print 2017 Aug. PMID 28775050
- [Result] Humbert M, Kovacs G, Hoeper MM, Badagliacca R, Berger RMF, Brida M, Carlsen J, Coats AJS, Escribano-Subias P, Ferrari P, Ferreira DS, Ghofrani HA, Giannakoulas G, Kiely DG, Mayer E, Meszaros G, Nagavci B, Olsson KM, Pepke-Zaba J, Quint JK, Radegran G, Simonneau G, Sitbon O, Tonia T, Toshner M, Vachiery JL, Vonk Noordegraaf A, Delcroix M, Rosenkranz S; ESC/ERS Scientific Document Group. 2022 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension. Eur Heart J. 2022 Oct 11;43(38):3618-3731. doi: 10.1093/eurheartj/ehac237. No abstract available. PMID 36017548